CLINICAL TRIAL: NCT05073120
Title: Survey Among Healthcare Professionals Treating Patients With Metastatic Breast Cancer in Selected European Countries to Evaluate Their Knowledge on Management of Hyperglycemia When Using Alpelisib
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CBYL719C2005
Record Dates: First submitted 2021-09-15; First posted 2021-10-11 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: educational material; PASS
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Piqray Prescriber's/HCP receiving the guide for hyperglycemia: HCPs prescribing Piqray in the EU/EEA provided with the Piqray Prescriber's/HCP Guide for hyperglycemia (educational material).
  Interventions: Other: Piqray Prescriber's/HCP guide for hyperglycemia

INTERVENTIONS:
Other: Piqray Prescriber's/HCP guide for hyperglycemia — oncologists/healthcare professionals (HCPs) prescribing Piqray in the EU/EEA were provided with the Piqray Prescriber's/HCP Guide for hyperglycemia (educational material). The educational material aimed to provide oncologists/HCPs prescribing Piqray with additional measures/guidance prior to, and during treatment with Piqray for the identification and management of hyperglycemia.

SUMMARY:
This was a multinational, non-interventional, cross-sectional survey conducted among HCPs based in the EU/EEA who prescribe Piqray. The survey assessed the knowledge of HCPs prescribing Piqray in relation to the management of hyperglycemia in patients treated with Piqray.

ELIGIBILITY:
Inclusion Criteria:

* Had prescribed Piqray to at least 1 locally advanced or MBC patient within 6 months prior to completing the survey.
* Provided permission to share their anonymized responses in aggregate with EMA or NCAs, if requested.

Exclusion Criteria:

HCPs who are direct employees of Novartis, the EMA (or any other regulatory bodies), or ICON.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oncologists/healthcare professionals (HCPs) prescribing Piqray in the EU/EEA provided with the Piqray Prescriber's/HCP Guide for hyperglycemia (educational material).
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
assess HCPs' knowledge and understanding of the key information included in the Piqray Prescriber's/HCP Guide for hyperglycemia | Throughout study completion, an average of 1 year
  The primary endpoint was a composite endpoint based on the percentages of HCPs with correct responses to all questions included in the composite regarding the below information:
  * Risk of hyperglycemia and its potential risk factors
  * Signs and symptoms of hyperglycemia
  * Recommendations for monitoring for hyperglycemia prior to, and during, treatment with Piqray
  * Recommendations for managing hyperglycemia during treatment with Piqray. Specifically, the primary endpoint was a weighted composite knowledge score aggregated across the following survey questions: 4A, 5A-C, 6, 8A-C, 10, and 12-15. It was calculated as the number of all correctly answered questions divided by the number of all answered questions (i.e. questions that were answered either correct and not correct - unanswered questions are excluded).

SECONDARY OUTCOMES:
Assess HCPs' reported levels of receipt, and reading, of the Piqray Prescriber's/HCP Guide for hyperglycemia | Throughout study completion, an average of 1 year
  Assessed as the percentages of HCPs who report receipt and reading of the same (survey questions 1, 2).
Assess HCPs' knowledge levels for each survey question regarding knowledge of, and management of, hyperglycemia | Throughout study completion, an average of 1 year
  Assessed as the percentages of HCPs with correct responses to each question (individual responses to survey questions 4-15).
Assess the primary source from which HCPs learned about the messages included in the Piqray Prescriber's/HCP Guide for hyperglycemia | Throughout study completion, an average of 1 year
  Assessed as the percentages of HCPs who report using each of the possible sources as the primary source they used (survey question 3).

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No